CLINICAL TRIAL: NCT06471491
Title: Driving Pressure-guided Positive End-expiratory Pressure to Prevent Postoperative Atelectasis in Obese Children: a Prospective, Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PEEP
Record Dates: First submitted 2024-05-31; First posted 2024-06-24 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Driving Pressure; Positive End-expiratory Pressure; Postoperative Atelectasis; Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung protective ventilation group (Experimental): PEEP was titrated individually in a sequential manner after mechanical ventilation. According to previous studies, PEEP was 5 cmH2O, inspiratory pressure was 20 cmH2O, and respiratory rate was set according to patient age. PEEP and inspiratory pressure were increased by 5 cmH2O every 30 seconds until PEEP was 15 cmH2O and inspiratory pressure 30 cmH2O. This was followed by a decreasing amplitude of 2 cmH2O to 3 cmH2O starting from 15 cmH2O, and each PEEP level was maintained for 4 to 5 respiratory cycles.The PEEP was at the lowest driving pressure was applied throughout the procedure. The PEEP level resulting in the lowest driving pressure was applied during surgery.
  Interventions: Other: Driving pressure-guided positive end-expiratory pressure
- Traditional mechanical ventilation group (No Intervention): In the traditional mechanical ventilation group, a fixed PEEP of 5 cm H2O was applied.

INTERVENTIONS:
Other: Driving pressure-guided positive end-expiratory pressure — Driving pressure-guided positive end-expiratory pressure during the surgical procedure
  Arms: Lung protective ventilation group

SUMMARY:
At present, the use of lung protective ventilation strategies in children is mainly based on adult and intensive care unit data. Although obese children may benefit more from lung protective ventilation, there are few studies on the use of lung protective ventilation strategies in obese children during surgery. Therefore, the investigators hypothesized that intraoperative use of LPV strategies in obese pediatric surgery patients can reduce atelectasis and improve the incidence of postoperative pulmonary complications.

DETAILED DESCRIPTION:
In the lung protective ventilation group, PEEP was titrated individually in a sequential manner after mechanical ventilation. According to previous studies, PEEP was 5 cmH2O, inspiratory pressure was 20 cmH2O, and respiratory rate was set according to patient age. PEEP and inspiratory pressure were increased by 5 cmH2O every 30 seconds until PEEP was 15 cmH2O and inspiratory pressure 30 cmH2O. This was followed by a decreasing amplitude of 2 cmH2O to 3 cmH2O starting from 15 cmH2O, and each PEEP level was maintained for 4 to 5 respiratory cycles.The PEEP was at the lowest driving pressure was applied throughout the procedure. The PEEP level resulting in the lowest driving pressure was applied during surgery. In the traditional mechanical ventilation group, a fixed PEEP of 5 cm H2O was applied. The investigators compared the incidence of postoperative atelectasis between the two groups using lung ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-18 years old;
* According to the People's Republic of China health industry standard "Overweight and Obesity Screening threshold for school-age children and adolescents WS_T586-2018" defined as obesity;
* American Society of Anesthesiologists (ASA) grades I - II;
* Children with healthy lungs and hearts;
* Patients with general anesthesia under tracheal intubation;
* Clear mind and able to cooperate with the anesthesiologist to receive treatment;
* Patients who plan to have elective surgery under general anesthesia and the estimated operation duration is ≥2 hours.

Exclusion Criteria:

* PEEP contraindications: (a) bronchopleural fistula; (b) hypovolemic shock; (c) right ventricular failure;
* American Society of Anesthesiologists (ASA) grade greater than II;
* Pulmonary dysfunction, congenital heart disease children;
* Refusal to participate in the study and/or use personal data, preoperative intubation or ventilation of children;
* Children with upper respiratory tract infection within 2 weeks.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of atelectasis in both groups at the end of surgery | at the end of surgery
  Incidence of atelectasis in both groups at the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhou, Study Chair — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No